CLINICAL TRIAL: NCT05996133
Title: Comparing Multifidus Cervicis Plane Block Vs. Sham Block, In Reducing Postoperative Pain And Opioid Consumption In Patients Undergoing Elective Primary Posterior Cervical Spine Fusion Surgery
Brief Title: Multifidus Cervicis Plane Block Vs. Sham Block For Posterior Cervical Spine Fusion Surgery
Acronym: MCP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Pranjali P Kainkaryam, MD, Director of Regional Anesthesia & Acute Pain Management, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HHC-2023-0156
Record Dates: First submitted 2023-07-26; First posted 2023-08-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spine Fusion
Keywords: Posterior cervical spine fusion surgery; Multifidus Cervicis Plane Block
MeSH Terms: conditions — Klippel-Feil Syndrome | interventions — Bupivacaine; Dexamethasone; Epinephrine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, double-blinded, randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: This is a double-blinded study, patients, research coordinators who collect data, spine surgeons, and other health care providers will all be blinded to the study group assignments to minimize bias and maximize the validity of study results. The block-performing anesthesiologists/investigators, the block nurse, and the senior scientist will not be blinded to the study group assignments.
  Patients will not be unblinded after they complete the study or during the study unless a participant experiences a serious adverse event that is unexpected and related to the study intervention (MCP or sham block) and the course of treatment needs to be adjusted. Unblinding in this situation will be the decision of the principal investigator (PI). The PI will contact the Senior Scientist to get the patient's group assignment, and the PI will then unblind the patient (i.e., tell the patient about the assigned group), and take any additional necessary course of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MCP Block (Experimental): Bilateral Multifidus Cervicis plane block using 30 mL of 0.25% bupivacaine + 0.5 mL (5 mg) preservative-free dexamethasone + 0.1 mL epinephrine 1:400,000.
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj
- Sham Block (Sham Comparator): Bilateral sham block using 3 mL of normal saline injections subcutaneously on the neck.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.25% Inj — 30 mL of 0.25% bupivacaine + 0.5 mL (5 mg) preservative-free dexamethasone + 0.1 mL epinephrine 1:400,000.
  Other Names: Dexamethasone; Epinephrine
  Arms: MCP Block
Other: Normal saline — 3 mL normal saline
  Arms: Sham Block

SUMMARY:
The goal of this randomized, double-blinded, clinical trial is to assess the benefit of administering a Multifidus Cervicis Plane (MCP) block compared to a sham block as a method of postoperative pain control in patients undergoing posterior cervical spine fusion surgery. The main question it aims to answer is if the MCP block group will have reduced maximum pain scores during the first 24 postoperative hours compared to the sham block group.

Participants will receive preoperative bilateral MCP blocks on the back of their neck using the standard of care local anesthetic solution that consists of 30 mLs 0.25% Bupivacaine + 0.5 mL (5 mg) preservative-free Dexamethasone + 0.1 mL Epinephrine (MCP block group). Researchers will compare the MCP block to the preoperative sham block which consists of injecting 3 mL of normal saline into the same area (Sham block group) to compare the postoperative pain scores between the groups as a main objective. The secondary objectives are:

* Postoperative opioid consumption during hospitalization and at 2 weeks after discharge.
* The amount and type of non-opioid analgesics used during hospitalization.
* The occurrence of postoperative nausea and vomiting (PONV) and the use of antiemetics.
* Hospital and Post Anesthesia Care Unit length of stay (LOS).
* Monitor the safety of the study interventions during hospitalization and readmissions within 30 days of discharge.
* Patient satisfaction with pain management and overall satisfaction with the surgery experience.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 40-80 years old, males and females, of any race and any ethnic group.
2. Patients are scheduled for elective primary posterior cervical spine fusion surgery (CSFS) to be performed by one of the spine surgeons in the study.
3. Ability to speak and read English
4. Patients with American Society of Anesthesiology (ASA) physical status score I- IV

Exclusion Criteria:

1. Emergency posterior CSFS.
2. Revision surgery or history of previous cervical spine surgery
3. History of allergy to local anesthetics or steroids.
4. Patients who are coagulopathic at the time of surgery
5. Patients with contraindications to MCP blocks, including but not limited to anatomical abnormality or previous surgical intervention that limits or prevents receiving the blocks
6. Infection at the site of the block.
7. Weight < 40 kg to avoid local anesthetic toxicity.
8. Patients on chronic or continuous opioid use of > 50 MME (morphine milli-equivalent) per day for at least 30 days within 90 days prior to surgery.
9. Patients with a history of chronic inflammatory conditions such as multiple sclerosis
10. Refusal to participate or lack of providing the study consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The maximum postoperative pain score | Up to 24 hours after surgery
  The maximum pain score for the past 24 postoperative hours, on a scale from 0-10 where 0 is no pain and 10 is severe pain reported by participants using the validated tool; Brief Pain Inventory-Short Form.

SECONDARY OUTCOMES:
The maximum, average, minimum, and current pain scores | 0-24 hours; 24-48 hours; 48-72 hours and at 2 weeks (+/- 7 days) after discharge via a phone call.
  The maximum, average, minimum, and current pain scores for the past 24 hours, on a scale from 0-10 where 0 is no pain and 10 is severe pain, reported by participants daily and up to 72 postoperative hours and at 2 weeks after discharge using the validated tool; Brief Pain Inventory-Short Form.
Total opioid consumption | at 6th, 12th, 24th, 48th, and 72nd postoperative hours, and at 2 weeks (+/- 7 days) after discharge.
  The total intraoperative and postoperative opioid consumption will be measured in morphine MilliEquivalent (MME) during hospitalization on the 6th, 12th, 24th, 48th, and 72nd postoperative hours, and at 2 weeks (+/- 7 days) after discharge via a phone call using a question asking if the patient is still using opioids (yes/no)
Non- opioid analgesics use | Up to 72 hours postoperative
  The number of non-opioid analgesics used (frequency), including NSAIDs, muscle relaxants, and gabapentin at any time throughout hospitalization up to 72 hours postoperatively.
Postoperative nausea/vomiting scores | Daily at 24th, 48th, and 72th postoperative hours
  Postoperative nausea/vomiting scores will be collected using the Simplified Postoperative Nausea and Vomiting Impact Scale, a validated measure that consists of two questions, each with a possible response score of 0-3. Response score totals of 0-2 require no intervention. Response score totals of 3-4 may necessitate antiemetic medication. Response score totals of 5-6 are considered clinically important nausea requiring medication intervention, as this would constitute patients with excessive vomiting.
Hospital and Post Anesthesia Care Unit length of stay | Up to 72 postoperative hours
  Hospital and PACU length of stay will be calculated in hours from the date and time of admission and discharge from the electronic medical records.
The occurrence of block complications | Up to 72 postoperative hours
  The occurrence of block complications will be collected during hospitalization will be assessed daily for up to the discharge from the hospital.
Participant satisfaction with the pain management service and the overall surgery experience | at 72nd postoperative hour and at 2 weeks (+/- 7 days) after discharge via a phone call
  Using the Customer Satisfaction Score (CSAT) tool, prior to discharge and at 2 weeks (+/- 7 days) after discharge via a phone call by the ARC. By asking participants to rate their satisfaction with pain management service and the overall surgery experience on a five-point scale: 1- very unsatisfied; 2- Unsatisfied; 3- Neutral; 4- Satisfied; and 5- Very satisfied. The metric will be looking specifically at the percentage of happy patients. The CSAT percentage score is calculated by looking at the 4 to 5 ratings. The formula is: (The total Number of 4 and 5 responses) ÷ (Number of total responses) x 100 = % of satisfied patients, a score of 80% will be considered 'good'.
Antiemetics used | up to 72 postoperative hours
  The number of doses (frequency) of intra and postoperative antiemetics will be collected up to 72 postop hours.

CONTACTS AND LOCATIONS:
Overall Officials: Pranjali Kainkaryam, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Minor PD, Macadam AJ, Stone DM, Almond JW. Genetic basis of attenuation of the Sabin oral poliovirus vaccines. Biologicals. 1993 Dec;21(4):357-63. doi: 10.1006/biol.1993.1096. No abstract available. PMID 8024751
- [Background] Youssef JA, Heiner AD, Montgomery JR, Tender GC, Lorio MP, Morreale JM, Phillips FM. Outcomes of posterior cervical fusion and decompression: a systematic review and meta-analysis. Spine J. 2019 Oct;19(10):1714-1729. doi: 10.1016/j.spinee.2019.04.019. Epub 2019 May 7. PMID 31075361
- [Background] Raja A, Patel P, Mesfin FB. Spinal Stenosis(Archived). 2023 Jun 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441989/ PMID 28723018
- [Background] Ohgoshi Y, Kurahashi K. Cervical interfascial plane (CIP) block and multifidus cervicis plane (MCP) block: Similarities and tips. J Clin Anesth. 2017 Sep;41:55. doi: 10.1016/j.jclinane.2017.06.014. Epub 2017 Jun 27. No abstract available. PMID 28802607
- [Background] Ohgoshi Y, Kubo EN. Inter-semispinal plane block for cervical spine surgery. J Clin Anesth. 2018 May;46:94-95. doi: 10.1016/j.jclinane.2018.02.007. Epub 2018 Feb 9. No abstract available. PMID 29433034
- [Background] Ahiskalioglu A, Yayik AM, Doymus O, Selvitopi K, Ahiskalioglu EO, Calikoglu C, Alici HA, Karaca O. Efficacy of ultrasound-guided modified thoracolumbar interfascial plane block for postoperative analgesia after spinal surgery: a randomized-controlled trial. Can J Anaesth. 2018 May;65(5):603-604. doi: 10.1007/s12630-018-1051-0. Epub 2018 Jan 9. No abstract available. PMID 29318534
- [Background] Mohamed, Z.E., Zarad, C.A., Flifel, M.E. et al. The efficacy of ultrasound-guided multifidus cervicis plane block versus greater occipital nerve block for cervicogenic headache. Egypt J Neurol Psychiatry Neurosurg 57, 11 (2021). https://doi.org/10.1186/s41983-020-00262-4
- [Background] Adamczyk K, Koszela K, Zaczynski A, Niedzwiecki M, Brzozowska-Mankowska S, Gasik R. Ultrasound-Guided Blocks for Spine Surgery: Part 1-Cervix. Int J Environ Res Public Health. 2023 Jan 23;20(3):2098. doi: 10.3390/ijerph20032098. PMID 36767465